CLINICAL TRIAL: NCT00779675
Title: Real-World Assessment of Long-Term Infliximab Therapy for Psoriasis
Brief Title: Assessment of Long-Term Infliximab for Psoriasis (P05319)
Acronym: REALITY
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05319; MK-2155-139 (Other: Merck Study Number)
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2012-10-29 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab 5 mg/kg
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab administered intravenously at a dose of 5 mg/kg body weight at Weeks 0, 2, 6 and then every 8 weeks (Weeks 14, 22, 30, 38, and 46 for the Treatment Period and Week 54, 62, 70, 78, 86, and 94 for the Extended Treatment Period) as per the product monograph (PM; Canada), summary of product characteristics (SPC; European Union), or local labeling (for all other countries).
  Other Names: Remicade; SCH 215596

SUMMARY:
This is a prospective Phase 4, open-label, non-randomized, observational, multi-center study of infliximab in participants with plaque-type psoriasis to assess the clinical response in real-world practice of long-term maintenance therapy with infliximab 5 mg/kg body weight in a psoriasis population, prescribed in a regimen in accordance with the product monograph (PM) for Canada, the approved summary sheet of product characteristics (SPC) for countries in the European Union (EU), or per label according to local guidelines for all other participating countries.

DETAILED DESCRIPTION:
This study will be conducted in two phases: the 50-week treatment period and the 48-week extended treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a diagnosis of plaque-type psoriasis
* Participant's physician must have decided, with the subject's consent, to start treatment with infliximab
* Participant must demonstrate willingness to participate in the study and agree with the procedures of the study by signing the written informed consent
* For inclusion into the extended treatment period, participant must have completed 50 weeks of infliximab treatment in the treatment period
* For inclusion into the extended treatment period, participant must be continuing treatment with intravenous infliximab
* For inclusion into the extended treatment period, participant must have an improvement in their PASI score of greater than or equal to 25% at the time of entry into to the extended treatment period

Exclusion Criteria:

For the Treatment Period

* Given the non-interventional nature of the study, no specific exclusion criteria will be applied to a participant so long as the participant is eligible for the trial (Inclusion Criteria). The treating physician is expected, as in normal clinical practice, to follow the PM (Canada), the approved SPC (EU), or local labeling (for all other participating countries) regarding contraindications and precautions

For the Extended Treatment Period

* Given the non-interventional nature of the study, no specific exclusion criteria will be applied to a participant so long as the participant is receiving infliximab treatment in accordance with the PM (Canada), the approved SPC (EU), or local labeling (for all other participating countries) regarding contraindications, precautions, dosing and frequency of administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with plaque-type psoriasis in which the treating physician has selected for treatment with infliximab, in accordance with local clinical practices, will be advised about this trial. It is highly recommended that 30% of the participants enrolled be naïve to previous biologic therapy. For example, if a site recruits 10 participants, 3 out of these 10 participants should be naïve to previous biologic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2012-08 (Actual)

REFERENCES:
- [Result] Shear NH, Hartmann M, Toledo-Bahena M, Katsambas A, Connors L, Chang Q, Yao R, Nograles K, Popmihajlov Z; REALITY investigators. Long-term efficacy and safety of infliximab maintenance therapy in patients with plaque-type psoriasis in real-world practice. Br J Dermatol. 2014 Sep;171(3):631-41. doi: 10.1111/bjd.13004. Epub 2014 Aug 13. PMID 24673357

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab 5 mg/kg: Infliximab administered intravenously at a dose of 5 mg/kg body weight at Weeks 0, 2, 6 and then every 8 weeks (Weeks 14, 22, 30, 38, and 46 for the Treatment Period and Week 54, 62, 70, 78, 86, and 94 for the Extended Treatment Period) as per the product monograph (PM; Canada), summary of product characteristics (SPC; European Union), or local labeling (for all other countries).
Period: Treatment Period
Arm/Group | Infliximab 5 mg/kg
Started | 660 (One of the 660 participants did not receive study treatment.)
Completed | 328
Not Completed | 332
Not completed — Adverse Event | 87
Not completed — Treatment Failure | 80
Not completed — Transferred to Another Study | 38
Not completed — Lost to Follow-up | 23
Not completed — Withdrawal by Subject | 46
Not completed — Protocol Violation | 54
Not completed — Did Not Meet Protocol Eligibility | 1
Not completed — Administrative | 3
Period: Extended Treatment Period
Arm/Group | Infliximab 5 mg/kg
Started | 193 (Clinical responders during the treatment period could enter the extended treatment period.)
Completed | 147
Not Completed | 46
Not completed — Reasons unrelated to study treatment | 9
Not completed — Protocol Violation | 13
Not completed — Adverse Event | 6
Not completed — Treatment Failure | 11
Not completed — Protocol defined clinical event | 1
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 660
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230
  Male | 430

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Psoriasis Area Sensitivity Index (PASI)-75 Response at Week 50
Description: Participant PASI scores were used to measure the severity and extent of psoriasis. Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness and scaling of the largest psoriatic area in that region; these 4 totals (totals ranging from 0 to 16) are then multiplied by the standardized percentage of total body area that each region represents (head = 0.1 of body surface area, trunk = 0.2 of body surface area, arms=0.3 of the body surface area, and legs = 0.4 of body surface area). An assessment is then made of the percentage of the area in that body region that is involved by the psoriatic lesions; this is expressed by a score from 0 (0% involved) to 6 (100% involved) and this score is multiplied by the subtotal of the total body area of that region; the four region scores are then added to produce the total PASI score. PASI-75 response was defined as >=75% improvement in overall PASI score when compared to baseline.
Time Frame: Week 50
Population: The Efficacy Population includes all participants with a baseline PASI score within 14 days of the time of the first infusion and at least one post-baseline PASI score.
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 521
Participants | 296

2. Secondary Outcome: Number of Participants With a PASI-90 Response at Week 50 Among Participants With a PASI-90 Response at Week 14
Description: Participant PASI scores were used to measure the severity and extent of psoriasis. Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness and scaling of the largest psoriatic area in that region; these 4 totals (totals ranging from 0 to 16) are then multiplied by the standardized percentage of total body area that each region represents (head = 0.1 of body surface area, trunk = 0.2 of body surface area, arms=0.3 of the body surface area, and legs = 0.4 of body surface area). An assessment is then made of the percentage of the area in that body region that is involved by the psoriatic lesions; this is expressed by a score from 0 (0% involved) to 6 (100% involved) and this score is multiplied by the subtotal of the total body area of that region; the four region scores are then added to produce the total PASI score. PASI-90 response was defined as >= 90% improvement when compared to baseline.
Time Frame: Week 50
Population: The population consists of all participants that achieved a PASI-90 response at treatment Week 14.
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 183
Participants | 104

3. Secondary Outcome: Number of Particpants With a PASI-90 or PASI-75 at Week 50 Among Participants With a PASI-75 Response at Week 14
Description: Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness and scaling of the largest psoriatic area in that region; these 4 totals (totals ranging from 0 to 16) are then multiplied by the standardized percentage of total body area that each region represents (head = 0.1 of body surface area, trunk = 0.2 of body surface area, arms=0.3 of the body surface area, and legs = 0.4 of body surface area). An assessment is then made of the percentage of the area in that body region that is involved by the psoriatic lesions; this is expressed by a score from 0 (0% involved) to 6 (100% involved) and this score is multiplied by the subtotal of the total body area of that region; the four region scores are then added to produce the total PASI score. PASI-90 and PASI-75 response were defined as >=90% improvement and a >=75% improvement, respectively, in overall PASI score when compared to baseline.
Time Frame: Week 50
Population: The population consists of all participants that achieved PASI-75 response by treatment Week 14.
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 317
Participants
  PASI-75 Response | 205
  PASI-90 Response | 152

4. Secondary Outcome: Number of Participants With a PASI-90, PASI-75, or PASI-50 Response at Week 50 Among Participants With a PASI-50 Response at Week 14
Description: Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness and scaling of the largest psoriatic area in that region; these 4 totals (ranging from 0 to 16) are then multiplied by the standardized percentage of total body area that each region represents (head = 0.1 of body surface area, trunk = 0.2 of body surface area, arms=0.3 of the body surface area, and legs = 0.4 of body surface area). An assessment is then made of the percentage of the area in that body region that is involved by the psoriatic lesions; this is expressed by a score from 0 (0% involved) to 6 (100% involved) and this score is multiplied by the subtotal of the total body area of that region; the four region scores are then added to produce the total PASI score. PASI-50, PASI-75, and PASI-90 response were defined as >=50%, >=75%, >=90% improvement in PASI score versus baseline.
Time Frame: Week 50
Population: The population includes all participants that achieved a PASI-50 response at treatment Week 14.
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 415
Participants
  PASI-50 Response | 292
  PASI-75 Response | 238
  PASI-90 Response | 170

5. Secondary Outcome: Number of Participants With a PASI-90 Response at Week 98 Among Participants With a PASI-90 Response at Week 50 and Who Entered the Extended Treatment Period
Description: Participant PSAI scores were used to measure the severity and extent of psoriasis. Using a scale of 0=none to 4=very severe, each body region (head, trunk, arms, and legs) is rate for redness, thickness and scaling of the largest psoriatic area in that region; these 4 totals (ranging from 0 to 16) are then multiplied by the standardized percentage of total body area that each regon represents (head=0.1 of body surface area, trunk=0.2 of body surface area, arms=0.3 of body surface area, legs=0.4 of body surface area). An assessment is then made of the percentage of the area in that body region that is involved by the psoriatic lesions; this is expressed by a score from 0 (0% involved) to 6 (100% involved) and this score is multipled by the subtotal of the body area of that region; the four region scores are then added to produce the total PASI score. PSAI-90 response was defined as >=90% improvement in overall PASI score when compared to baseline.
Time Frame: Week 98
Population: The population consists of all participants that achieved PASI-90 response at Week 50 and entered the extended treatment phase.
Measure: Number; unit: Participants
Groups:
- Infliximab 5 mg/kg: Infliximab administered intravenously at a dose of 5 mg/kg body weight at Weeks 0, 2, 6 and then every 8 weeks (Weeks 14, 22, 30, 38, and 46 for the Treatment Period and Week 54, 62, 70, 78, 86, and 94 for the Extended Treatment Period) as per the product monograph (PM; Canada), summary of product characteristics (SPC; European Union), or local labelling (for all other Countries).
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 106
Participants | 66

6. Secondary Outcome: Number of Participants With a PASI-90, PASI-75, or PASI-50 Response at Week 98 Among Participants With a PASI-50 Response at Week 50 and Who Entered the Extended Treatment Period
Description: Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness and scaling of the largest psoriatic area in that region; these 4 totals (ranging from 0 to 16) are then multiplied by the standardized percentage of total body area that each region represents (head = 0.1 of body surface area, trunk = 0.2 of body surface area, arms=0.3 of the body surface area, and legs = 0.4 of body surface area). An assessment is then made of the percentage of the area in that body region that is involved by the psoriatic lesions; this is expressed by a score from 0 (0% involved) to 6 (100% involved) and this score is multiplied by the subtotal of the total body area of that region; the four region scores are then added to produce the total PASI score. PASI-50, PASI-75, and PASI-90 response were defined as >=50%, >=75%, >=90% improvement in PASI score versus baseline, respectively.
Time Frame: Week 98
Population: The population includes all participants that achieved PASI-50 response at Week 50 and entered the extended treatment phase.
Measure: Number; unit: Participants
Groups:
- Infliximab 5 mg/kg: Infliximab administered intravenously at a dose of 5 mg/kg body weight at Weeks 0, 2,6, and then every 8 weeks (Weeks 14, 22, 30, 38, and 46 for the Treatment Period and Weeks 54, 62, 70, 78, 86, and 94 for the Extended Treatment Period) as per the product monograph (PM; Canada), summary of product characteristics (SPC; European Union), or local labelling (for all other Countries)
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 158
Participants
  PASI-90 | 81
  PASI-75 | 107
  PASI-50 | 122

7. Secondary Outcome: Change From Baseline in Mean PASI Score
Description: Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness and scaling of the largest psoriatic area in that region; these 4 totals (ranging from 0 to 16) are then multiplied by the standardized percentage of total body area that each region represents (head = 0.1 of body surface area, trunk = 0.2 of body surface area, arms=0.3 of the body surface area, and legs = 0.4 of body surface area). An assessment is then made of the percentage of the area in that body region that is involved by the psoriatic lesions; this is expressed by a score from 0 (0% involved) to 6 (100% involved) and this score is multiplied by the subtotal of the total body area of that region; the four region scores are then added to produce the total PASI score. Decreasing scores are indicative of improvement in overall PASI score.
Time Frame: Baseline, Week 14, Week 30, Week 50, Week 62, Week 78, Week 98
Population: The population consists of all participants with a baseline PASI score and a subsequent score at Week 14, 30, 50, 62, 78,and 98.
Measure: Mean (95% Confidence Interval); unit: Score on a Scale
Groups:
- Infliximab 5 mg/kg: Infliximab administered intravenously at a dose of 5 mg/kg of body weight at Week 0, 2, 6 and then every 8 weeks (Weeks 14, 22, 30, 38, and 46 for the Treatment Period and Weeks 54, 62, 70, 78, 86, and 94 for the Extended Treatment Period) as per the product monograph (PM; Canada), summary of product characterisitics (SPC; European Union), or local labelling (for all other countries).
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 169
Score on a Scale
  Week 14 (n=166) | -17.3 (-17.3) [-18.87 to -15.71]
  Week 30 (n=165) | -18.0 (-18.0) [-19.66 to -16.38]
  Week 50 (n=165) | -18.4 (-18.4) [-20.01 to -16.74]
  Week 62 (n=136) | -17.8 (-17.8) [-19.67 to -15.98]
  Week 78 (n=143) | -17.5 (-17.5) [-19.22 to -15.70]
  Week 98 (n=142) | -17.3 (-17.3) [-19.06 to -15.55]

8. Secondary Outcome: Number of Participants With a PASI-90 or PASI-75 Response at Week 98 Among Participants Who Had a PASI-75 Response at Week 50 and Who Entered the Extended Treatment Phase
Description: PASI socres were used to measure the severity and extent of psoriasis. Using a scale of 0=nonoe to 4=very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness, and scaling of the largest psoriatic area in that region; thse 4 totals (ranging from 0 to 16) are then multipled by the standardized percentage of total body area that region represents (head=0.1 of body surface area, trunk=0.2 of body surface area, arms=0.3 of body surface area, and legs=0.4 of body surface area). An assessment is then made of the percentage of area in that body region that is involved by the psoriatic lesions; this is expressed by a score from 0 (0% involved) to 6 (100% involved) and this score is multiplied by the subtotal of the total body area of that region; the four region scores are then added to produce the total PASI score. PASI-90 and PASI-75 response were defined at >=90% and >=75% improvement in overall PASI score when compared to baselne, respectively.
Time Frame: Week 98
Population: The population consisted of participants who were in the efficacy population of the treatment phase and who entered into the extended treatment phase and had a PASI-75 response at Week 50 with at least one PASI evaluation during the extended treatment phase.
Measure: Number; unit: Participants
Groups:
- Infliximab 5 mg/kg: Infliximab administered intravenously at a dose of 5 mg/kg of body weight at Weeks 0, 2, 6, and then every 8 weeks (Week 14, 22, 30, 38, and 46 for the Treatment Period and Weeks 54, 62, 70, 78, 86, and 94 for the Extended Treatment Period) as per the product monograph (PM; Canada, summary of product characteristics (SPC; European Union), or local labelling (for all other countries).
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 141
Participants
  PASI-90 | 77
  PASI-75 | 101

9. Secondary Outcome: Change From Baseline in Mean Dermatology Life Quality Index (DLQI)
Description: The DLQI assesses the impact of psoriasis on the participants's daily life. DLQI total score comprises 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. DLQI total scores range from 0 to 30, with 0 corresponding to the best quality of life and 30 to the worst with 0-1=no effect on the partipant's life, 2-5=small effect on the participant's life, 6-10= moderate effect on the participant's life, 11=20= very large effect on participant's life, and 21-30 = extremely large effect on participant's life.
Time Frame: Baseline, Week 50, Week 62, Week 78, Week 98
Population: The population consisted of all participants with a DLQI measurement at baseline and at each time point.
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 169
Score on a Scale
  Week 50 (n=149) | 9.8 (0.61) [-10.98 to -8.56]
  Week 62 (n=131) | 9.0 (0.77) [-10.54 to -7.49]
  Week 78 (n=134) | 9.7 (0.69) [-11.07 to -8.32]
  Week 98 (n=140) | 9.4 (0.70) [-10.78 to -7.99]

10. Secondary Outcome: Number of Participants With A DLQI Score of 0 or 1 in the Extended Treatment Phase
Description: as for outcome 9
Time Frame: Week 50, Week 62, Week 78, Week 98
Population: The population consisted of all participants with a DLQI measurement at each time point.
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 169
Participants
  Week 50, DLQI=0 | 77
  Week 50, DLQI=0 or 1 | 102
  Week 50, DLQI >1 | 51
  Week 50, DLQI Missing | 16
  Week 62, DLQI=0 | 51
  Week 62, DLQI=0 or 1 | 75
  Week 62, DLQI >1 | 57
  Week 62, DLQI Missing | 37
  Week 78, DLQI=0 | 57
  Week 78, DLQI=0 or 1 | 80
  Week 78, DLQI >1 | 55
  Week 78, DLQI Missing | 34
  Week 98, DLQI=0 | 67
  Week 98. DLQI=0 or 1 | 84
  Week 98, DLQI >1 | 57
  Week 98, DLQI Missing | 28

11. Secondary Outcome: Number of Participants With a PASI-50, PASI-75, PASI-90, or PASI-100 Response at Week 98
Description: Using a scale of 0=none to 4= very severe, each body region (head, trunk, arms, and legs) is rated for redness, thickness and scaling of the largest psoriatic area in that region; these 4 totals (ranging from 0 to 16) are then multiplied by the standardized percentage of total body area that each region represents (head = 0.1 of body surface area, trunk = 0.2 of body surface area, arms=0.3 of the body surface area, and legs = 0.4 of body surface area). An assessment is then made of the percentage of the area in that body region that is involved by the psoriatic lesions; this is expressed by a score from 0 (0% involved) to 6 (100% involved) and this score is multiplied by the subtotal of the total body area of that region; the four region scores are then added to produce the total PASI score. PASI-50, PASI-75, PASI-90, and PASI-100 response were defined as >=25%, >=50%, >=75%, >=90%, =100% improvement in PASI score versus baseline, respectively.
Time Frame: Week 98
Population: The population consisted of participants who were in the efficacy population of the treatment phase and who entered into the extended treatment phase with at least one PASI evaluation during the extended treatment phase.
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 169
Participants
  PASI-50 | 129
  PASI-75 | 112
  PASI-90 | 82
  PASI-100 | 35

12. Secondary Outcome: Number of Participants Who Achieved a PASI-75 Response at Week 50 by Age
Description: as for outcome 1
Time Frame: Week 50
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 521
Participants
  Age <65 years (n=469) | 264
  Age >=65 years (n=52) | 32

13. Secondary Outcome: Number of Participants Who Achieved a PASI-75 Response at Week 50 by Gender
Description: as for outcome 1
Time Frame: Week 50
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 521
Participants
  Male (n=344) | 199
  Female (n=177) | 97

14. Secondary Outcome: Number of Participants Who Achieved a PASI-75 Response at Week 50 by Race
Description: as for outcome 1
Time Frame: Week 50
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 521
Participants
  Caucasian (n=436) | 235
  Non-Caucasian (n=85) | 61

15. Secondary Outcome: Number of Participants Who Achieved a PASI-75 Response at Week 50 by the Presence of Nail Psoriasis at Baseline
Description: as for outcome 1
Time Frame: Week 50
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 521
Participants
  Nail Psoriasis Present at Baseline (n=308) | 171
  Nail Psoriasis Absent at Baseline (n=213) | 125

16. Secondary Outcome: Number of Participants Who Achieved a PASI-75 Response at Week 50 by PASI Score at Baseline
Description: as for outcome 1
Time Frame: Week 50
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab 5 mg/kg
Number analyzed (Participants) | 521
Participants
  Baseline PASI <12 (n=167) | 77
  Baseline PASI >=12 (n=354) | 219

ADVERSE EVENTS:
Time Frame: Up to Week 98
Arm/Group | Infliximab 5 mg/kg
Serious Adverse Events (participants affected / at risk) | 56/659
Other Adverse Events (participants affected / at risk) | 0/659
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab 5 mg/kg (N=659)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1)
Coronary Artery Stenosis (Cardiac disorders) | 1 (1)
Left Ventricular Failure (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1)
Drug Interaction (General disorders) | 1 (1)
Cytolytic Hepatitis (Hepatobiliary disorders) | 2 (2)
Gallbladder Polyp (Hepatobiliary disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Clostridial Infection (Infections and infestations) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis Salmonella (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Lymph Node Tuberculosis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Tuberculosis (Infections and infestations) | 2 (2)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (2)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 1 (1)
Tuberculin Test Positive (Investigations) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (2)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Malignant Peritoneal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal Ganglia Haemorrhage (Nervous system disorders) | 1 (1)
Intraventricular Haemorrhage (Nervous system disorders) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Enuresis (Renal and urinary disorders) | 1 (1)
Renal Colic (Renal and urinary disorders) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Generalised Exanthematous Pustulosis (Skin and subcutaneous tissue disorders) | 2 (2)
Erythrodermic Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3)
Pregnancy of Partner (Social circumstances) | 1 (1)
Inguinal Hernia Repair (Surgical and medical procedures) | 1 (1)
Umbilical Hernia Repair (Surgical and medical procedures) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1)
Liver Function Test Abnormal (Investigations) | 1 (1)
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder Tamponade (Renal and urinary disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Hip Arthroplasty (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data.